CLINICAL TRIAL: NCT02806414
Title: A Single Site Evaluation of the Inhibitory Effects of Topical Ivermectin on Serine Protease Activity and Production of LL-37 Cathelicidin Peptide, Biochemical Markers of Rosacea-specific Inflammation and on the Skin Microbiome in Rosacea.
Brief Title: Evaluation of the Inhibitory Effects of Topical Ivermectin on Markers of Rosacea Specific Inflammation.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Tissa Hata, MD, Professor of Dermatology, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD 160765
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ivermectin (Experimental): All subjects will be treated with topical ivermectin daily for up to 12 weeks.
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin
  Other Names: Soolantra

SUMMARY:
This study will assess the role of topical Ivermectin 1% cream and its effect on protease and antimicrobial peptide expression and on the skin microbiome (the microorganisms that live on the skin) in rosacea. This is a single-site 16-week open-label study at University of California, San Diego. The investigators will do this by first measuring serine protease activity and cathelicidin and skin microbiome of all subjects. All subjects will receive Ivermectin topical cream and will be instructed on how to apply it daily for 12 weeks. Participants will return for monthly visits during which their clinical symptoms of facial redness and number of facial papules will be scored, and they will have repeat tape stripping and/or skin swabs. At the end of the study, tape strips and skin swabs will be analyzed to determine serine protease activity and skin microbiome of participants at each of their visits and expression of cathelicidin (LL-37) mRNA. The investigators will then look at changes in serine protease activity and LL-37 expression and skin microbiome over time, and they will also determine whether or not these changes correlate with disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or non-pregnant female, 18 - 70 years of age.
* Subjects willing and able to give informed consent.
* Subjects willing and able to comply with the requirements of the study.
* Subject has the clinical diagnosis of rosacea with at least one inflammatory papule and at least mild erythema.
* Subject has been on a stable dose for greater than 3 months of medications for treatment of concurrent medical condition (including oral contraceptive pills, vasodilators, adrenergic blocking agents) OR the investigator has determined that the medications are unlikely to affect the patient's rosacea and/or treatment during the study
* Subject is in general good health in the opinion of the investigator.
* Subject has normal baseline labs or in the opinion of the investigator are values are not clinically significant and would not inhibit the ability to monitor the patient for both safety and efficacy throughout the study.

Exclusion Criteria:

* Subject has a diagnosis of Steroid Rosacea or Pyoderma Faciale (rosacea fulminans).
* Subject has used facial topical therapies (OTC drug products or prescription products) for any reason within the prior 28 days
* Subject has used systemic corticosteroid or systemic antibiotics (especially doxycycline, minocycline, tetracycline, metronidazole) within the prior 28 days.
* Subject has had laser or light-based treatment for rosacea within the prior 3 months.
* Subject has had systemic retinoids and retinoid derivatives over the past 6 months
* Subject has a known hypersensitivity or allergy to topical ivermectin or components of the vehicle.
* Subject is pregnant or lactating or planning a pregnancy during the duration of the study
* Subject has been treated with another investigational device or drug within 28 days prior to study enrollment or intends to participate in a clinical trial concurrent with this study
* Subject has clinically significant findings, medical history or conditions (other than rosacea), which in the opinion of the Investigator may compromise the study, treatment protocol, or safety of the patient or treatment allocation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tissa Hata, MD, Principal Investigator — UCSD Division of Dermatology
Locations (1):
- UCSD Division of Dermatology, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ivermectin: All subjects will be treated with topical ivermectin daily for up to 12 weeks.
  Ivermectin
Period: Overall Study
Arm/Group | Ivermectin
Started | 25
Completed | 23
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ivermectin
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Relative Trypsin-like Enzyme Activity
Description: Activity was quantified using a protease activity assay involving aprotinin, a known selective inhibitor of trypsin-related enzyme activity
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Ivermectin
Number analyzed (Participants) | 23
percentage of baseline | 1.10 [0.58 to 1.4]

2. Secondary Outcome: Relative Fold Change in Cathelicidin mRNA
Description: Ratio of fold change in cathelicidin mRNA at 12 weeks to fold change in cathelicidin mRNA at baseline
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: ratio
Arm/Group | Ivermectin
Number analyzed (Participants) | 11
ratio | 3.25 [.54 to 4.89]

ADVERSE EVENTS:
Time Frame: Baseline visit to follow-up phone visit (4 months total)
Arm/Group | Ivermectin
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 3/25
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin (N=25)
melanoma excision (Skin and subcutaneous tissue disorders) | 1 (1)
cold (Infections and infestations) | 1 (1)
mild bleeding (Investigations) | 1 (1) — intermittently from tape stripping site for 2 days
ear infection (Infections and infestations) | 1 (1)
epidermal inclusion cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT02806414/Prot_SAP_001.pdf